CLINICAL TRIAL: NCT05525910
Title: A Phase 1, Open-Label, Randomized, Single Dose, Crossover Study to Estimate the Relative Bioavailability of Nirmatrelvir and Ritonavir Following Oral Administration of 4 Different Fixed Dose Combination Tablet Formulations Relative to The Commercial Tablet Formulation in Healthy Adult Participants Under Fasted Conditions
Brief Title: Relative Bioavailability Study of Nirmatrelvir/Ritonavir 4 Different Fixed Dose Combination Tablets Relative to the Commercial Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671023
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Biological Availability; Healthy Participants
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nirmatrelvir; Paxlovid
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: Nirmatrelvir/ritonavir (Active Comparator): Nirmatrelvir and ritonavir tablets
  Interventions: Drug: Nirmatrelvir/ ritonavir
- Treatment B: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir test tablets
  Interventions: Drug: Nirmatrelvir/ritonavir
- Treatment C: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir test tablets
  Interventions: Drug: Nirmatrelvir/ritonavir
- Treatment D: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir test tablets
  Interventions: Drug: Nirmatrelvir/ ritonavir
- Treatment E: Nirmatrelvir/ ritonavir (Experimental): Nirmatrelvir/ ritonavir test tablets
  Interventions: Drug: Nirmatrelvir/ ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/ ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment A: Nirmatrelvir/ritonavir
Drug: Nirmatrelvir/ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment B: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment C: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/ ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment D: Nirmatrelvir/ ritonavir
Drug: Nirmatrelvir/ ritonavir — Single oral dose of nirmatrelvir/ritonavir tablets under fasted condition
  Arms: Treatment E: Nirmatrelvir/ ritonavir

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of nirmatrelvir/ritonavir of 4 different FDC tablet formulations relative to the commercial tablet formulation under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination (PE), laboratory tests, vital signs and standard 12 lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671023

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants were randomized and assigned to receive the study intervention.
Groups:
- Sequence 1: Treatment A-> B-> C-> D: Period 1: Treatment A: Single oral dose of nirmatrelvir/ritonavir 300 (2*150)/100 mg commercial tablets under fasted conditions (Reference).
  Period 2: Treatment B: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) fixed dose combination (FDC) tablets Test formulation 1 (low disintegrant) under fasted conditions (Test 1).
  Period 3: Treatment C: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 2 (high disintegrant) under fasted conditions (Test 2).
  Period 4: Treatment D: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 3 (high drug loading [HDL]) under fasted conditions (Test 3).
  Each enrolled participant participated in 4 study periods to receive 4 different treatments according to the sequence determined by randomization. On Day 1 of each period, participants received a single oral dose of treatment as per the randomization schedule and a minimum of 4 days washout was planned between each treatment.
- Sequence 2: Treatment B-> C-> D-> E: Period 1: Treatment B: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 1 (low disintegrant) under fasted conditions (Test 1).
  Period 2: Treatment C: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 2 (high disintegrant) under fasted conditions (Test 2).
  Period 3: Treatment D: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2* [150/50 mg]) FDC tablets Test formulation 3 (HDL) under fasted conditions (Test 3).
  Period 4: Treatment E: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (3*[100/33.3 mg]) FDC tablets Test formulation 4 under fasted conditions (Test 4).
  Each enrolled participant participated in 4 study periods to receive 4 different treatments according to the sequence determined by randomization. On Day 1 of each period, participants received a single oral dose of treatment as per the randomization schedule and a minimum of 4 days washout was planned between each treatment.
- Sequence 3: Treatment C-> D-> E-> A: Period 1: Treatment C: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 2 (high disintegrant) under fasted conditions (Test 2).
  Period 2: Treatment D: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 3 (HDL) under fasted conditions (Test 3).
  Period 3: Treatment E: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (3*[100/33.3 mg]) FDC tablets Test formulation 4 under fasted conditions (Test 4).
  Period 4: Treatment A: Single oral dose of nirmatrelvir/ritonavir 300 (2*150)/100 mg commercial tablets under fasted conditions (Reference).
  Each enrolled participant participated in 4 study periods to receive 4 different treatments according to the sequence determined by randomization. On Day 1 of each period, participants received a single oral dose of treatment as per the randomization schedule and a minimum of 4 days washout was planned between each treatment.
- Sequence 4: Treatment D-> E-> A-> B: Period 1: Treatment D: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 3 (HDL) under fasted conditions (Test 3).
  Period 2: Treatment E: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (3*[100/33.3 mg]) FDC tablets Test formulation 4 under fasted conditions (Test 4).
  Period 3: Treatment A: Single oral dose of nirmatrelvir/ritonavir 300 (2*150)/100 mg commercial tablets under fasted conditions (Reference).
  Period 4: Treatment B: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 1 (low disintegrant) under fasted conditions (Test 1).
  Each enrolled participant participated in 4 study periods to receive 4 different treatments according to the sequence determined by randomization. On Day 1 of each period, participants received a single oral dose of treatment as per the randomization schedule and a minimum of 4 days washout was planned between each treatment.
- Sequence 5: Treatment E-> A-> B-> C: Period 1: Treatment E: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (3*[100/33.3 mg]) FDC tablets Test formulation 4 under fasted conditions (Test 4).
  Period 2: Treatment A: Single oral dose of nirmatrelvir/ritonavir 300 (2*150)/100 mg commercial tablets under fasted conditions (Reference).
  Period 3: Treatment B: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 1 (low disintegrant) under fasted conditions (Test 1).
  Period 4: Treatment C: Single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 2 (high disintegrant) under fasted conditions (Test 2).
  Each enrolled participant participated in 4 study periods to receive 4 different treatments according to the sequence determined by randomization. On Day 1 of each period, participants received a single oral dose of treatment as per the randomization schedule and a minimum of 4 days washout was planned between each treatment.
Period: Period 1
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> C-> D-> E | Sequence 3: Treatment C-> D-> E-> A | Sequence 4: Treatment D-> E-> A-> B | Sequence 5: Treatment E-> A-> B-> C
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> C-> D-> E | Sequence 3: Treatment C-> D-> E-> A | Sequence 4: Treatment D-> E-> A-> B | Sequence 5: Treatment E-> A-> B-> C
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> C-> D-> E | Sequence 3: Treatment C-> D-> E-> A | Sequence 4: Treatment D-> E-> A-> B | Sequence 5: Treatment E-> A-> B-> C
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> C-> D-> E | Sequence 3: Treatment C-> D-> E-> A | Sequence 4: Treatment D-> E-> A-> B | Sequence 5: Treatment E-> A-> B-> C
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Per sponsor due to study timelines | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Treatment A-> B-> C-> D | Sequence 2: Treatment B-> C-> D-> E | Sequence 3: Treatment C-> D-> E-> A | Sequence 4: Treatment D-> E-> A-> B | Sequence 5: Treatment E-> A-> B-> C | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.3 (2.52) | 56.7 (4.16) | 50.0 (10.58) | 53.3 (17.10) | 51.7 (6.51) | 48.4 (12.64)
Age, Customized [Number; unit: Participants]
  18-44 years | 3 | 0 | 1 | 1 | 0 | 5
  45-64 years | 0 | 3 | 2 | 1 | 3 | 9
  >=65 years | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 0 | 2
  Male | 3 | 2 | 2 | 3 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 2 | 2 | 2 | 1 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 1 | 2 | 6
  White | 0 | 2 | 3 | 2 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCinf of Nirmatrelvir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time. AUCinf for nirmatrelvir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Nirmatrelvir/Ritonavir 300(2*150)/100 mg: Participants received a single oral dose of nirmatrelvir/ritonavir 300 (2*150)/100 mg commercial tablets under fasted conditions (Reference) on Day 1 of each treatment period.
- Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant: Participants received a single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 1 (low disintegrant) under fasted conditions (Test 1) on Day 1 of each treatment period.
- Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant: Participants received a single oral dose of nirmatrelvir/ritonavir 300/100 mg (2*[150/50 mg]) FDC tablets Test formulation 2 (high disintegrant) under fasted conditions (Test 2) on Day 1 of each treatment period.
- Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL: Participants received a single oral dose of nirmatrelvir/ritonavir 300/100 mg (2* [150/50 mg]) FDC tablets Test formulation 3 (HDL) under fasted conditions (Test 3) on Day 1 of each treatment period.
- Nirmatrelvir/Ritonavir 3*(100/33.3 mg): Participants received a single oral dose of nirmatrelvir/ritonavir 300/100 mg (3*[100/33.3 mg]) FDC tablets Test formulation 4 under fasted conditions (Test 4) on Day 1 of each treatment period.
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 27040 (36) | 29350 (28) | 30680 (21) | 28200 (40) | 33660 (29)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — Analysis done using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Ratio and 90% CI are expressed as percentages; Ratio (%) of Adjusted Geometric Means = 105.03, 90% CI 2-sided [94.54 to 116.68]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 109.15, 90% CI 2-sided [98.08 to 121.47]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 100.72, 90% CI 2-sided [90.79 to 111.74]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 110.45, 90% CI 2-sided [99.58 to 122.52]

2. Primary Outcome: AUClast of Nirmatrelvir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast). AUClast for nirmatrelvir was calculated by Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
ng*hr/mL | 26620 (37) | 28890 (28) | 30350 (21) | 27630 (42) | 33060 (31)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 104.86, 90% CI 2-sided [93.78 to 117.24]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 109.70, 90% CI 2-sided [97.93 to 122.89]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 100.14, 90% CI 2-sided [89.69 to 111.80]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 109.80, 90% CI 2-sided [98.36 to 122.57]

3. Primary Outcome: Cmax of Nirmatrelvir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: Cmax was defined as maximum plasma concentration. Cmax for nirmatrelvir was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
nanogram per milliliter (ng/mL) | 2709 (47) | 3111 (34) | 3181 (24) | 3051 (42) | 3556 (41)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 109.85, 90% CI 2-sided [94.97 to 127.06]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 114.69, 90% CI 2-sided [98.92 to 132.98]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 109.26, 90% CI 2-sided [94.64 to 126.14]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 115.98, 90% CI 2-sided [100.48 to 133.87]

4. Primary Outcome: AUCinf of Ritonavir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time. AUCinf for ritonavir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
ng*hr/mL | 3420 (76) | 3230 (81) | 3453 (54) | 2921 (85) | 4130 (62)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 88.85, 90% CI 2-sided [76.24 to 103.53]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 95.11, 90% CI 2-sided [81.41 to 111.11]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 85.74, 90% CI 2-sided [73.73 to 99.70]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 93.12, 90% CI 2-sided [80.09 to 108.26]

5. Primary Outcome: AUClast of Ritonavir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast). AUClast for ritonavir was calculated by Linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
ng*hr/mL | 3224 (76) | 3044 (84) | 3297 (53) | 2735 (87) | 3821 (66)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 88.43, 90% CI 2-sided [74.64 to 104.78]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 96.00, 90% CI 2-sided [80.80 to 114.06]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 84.11, 90% CI 2-sided [71.15 to 99.43]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 90.99, 90% CI 2-sided [76.99 to 107.54]

6. Primary Outcome: Cmax of Ritonavir Following the Administration of 4 Different Nirmatrelvir/Ritonavir FDC Tablets (Test Formulations) Compared to the Nirmatrelvir/Ritonavir 300(2*150)/100 mg Tablets (Reference Formulation)
Description: Cmax was defined as maximum plasma concentration. Cmax for ritonavir was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 1 of each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
ng/mL | 371.3 (67) | 334.2 (93) | 374.5 (47) | 319.5 (84) | 411.3 (77)
Statistical Analysis 1: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) Low Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 82.65, 90% CI 2-sided [65.85 to 103.74]
Statistical Analysis 2: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) High Disintegrant; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 94.85, 90% CI 2-sided [75.28 to 119.49]
Statistical Analysis 3: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL; Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 2*(150/50 mg) HDL; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 81.56, 90% CI 2-sided [65.18 to 102.07]
Statistical Analysis 4: Comparison: Nirmatrelvir/Ritonavir 300(2*150)/100 mg vs Nirmatrelvir/Ritonavir 3*(100/33.3 mg); Reference: Nirmatrelvir/ritonavir 300(2*150)/100 mg Test: Nirmatrelvir/ritonavir 3*(100/33.3 mg); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 88.38, 90% CI 2-sided [70.65 to 110.57]

7. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study treatment and up to approximately 51 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study treatment up to 35 days after last dose of study treatment (ie, up to 51 days)
Population: All participants who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
Participants
  Number of participants with all-causality TEAEs | 2 | 0 | 2 | 1 | 2
  Number of participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0
  Number of participants with treatment-related TEAEs | 0 | 0 | 0 | 0 | 0
  Number of participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Hematology, Chemistry, and Urinalysis
Description: Hematology included hemoglobin, hematocrit, red blood cell, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, etc. Chemistry included blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, fibrinogen, etc. Urinalysis included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy and culture. Clinical significance was judged by the investigator and those met the criteria of AE are listed here. Clinically significant laboratory abnormalities reported for at least 1 participant in the whole study are presented here. Baseline was defined as the last measurement taken prior to first dosing (Period 1 Day -1).
Time Frame: From baseline up to Day 4 of Period 4 (approximately 17 days)
Population: Participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 5
Participants
  Neutrophils (10^9/L) <0.8*lower limit of normal (LLN) | 0 | 0 | 0 | 1 | 0
  Monocytes/Leukocytes (%) >1.2*upper limit of normal (ULN) | 0 | 0 | 0 | 1 | 2
  Fibrinogen (mg/dL) >1.25*baseline: number analyzed (Participants) | 3 | 3 | 2 | 4 | 4
  Fibrinogen (mg/dL) >1.25*baseline | 2 | 0 | 0 | 1 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs (temperature, pulse rate and blood pressure) were obtained with participants following at least 5 minutes of supine rest. Clinical significance of vital signs was determined at the investigator's discretion. Baseline was defined as pre-dose measurement taken on Day 1 of each period.
Time Frame: From baseline up to Day 4 of Period 4 (approximately 16 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Values
Description: A complete physical examination (PE) included, at a minimum, height, weight, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief PE included, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant-reported symptoms. Clinical significance of physical examination values was determined at the investigator's discretion.
Time Frame: From baseline up to 35 days after last dose of study treatment (ie, up to 51 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG)
Description: A 12-lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured pulse rate, QT, and QTc intervals and QRS complex. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position. Clinical significance of ECG values was determined at the investigator's discretion. Baseline was defined as pre-dose measurement taken on Day 1 of Period 1.
Time Frame: From baseline up to Day 4 of Period 4 (approximately 16 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to 35 days after last dose of study treatment (ie, up to 51 days)
Arm/Group | Nirmatrelvir/Ritonavir 300(2*150)/100 mg | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL | Nirmatrelvir/Ritonavir 3*(100/33.3 mg)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 0/11 | 2/11 | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir/Ritonavir 300(2*150)/100 mg (N=11) | Nirmatrelvir/Ritonavir 2*(150/50 mg) Low Disintegrant (N=11) | Nirmatrelvir/Ritonavir 2*(150/50 mg) High Disintegrant (N=11) | Nirmatrelvir/Ritonavir 2*(150/50 mg) HDL (N=12) | Nirmatrelvir/Ritonavir 3*(100/33.3 mg) (N=12)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT05525910/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT05525910/SAP_001.pdf